CLINICAL TRIAL: NCT04480723
Title: A Prospective Multicenter Study for the Assessment of Biomarker Signatures for the Diagnosis of Pulmonary Hypertension (PH) in Patients at Low or Intermediate Probability of PH Undergoing Cardiac Magnetic Resonance Imaging (MRI) CIPHER-MRI
Brief Title: A Study for the Identification of Biomarker Signatures for Diagnosis of Pulmonary Hypertension (PH) in Participants at Low or Intermediate Probability of PH Undergoing Cardiac Magnetic Resonance Imaging
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR108827; NAPUH0003 (Other: Actelion)
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Low or Intermediate Probability of PH (Other): Participants who underwent a work-up for the suspicion of PH that includes transthoracic echocardiography (TTE) and who were considered to have a low or intermediate probability of PH according to TTE (local interpretation) will be enrolled. Blood samples will be taken and a cardiac magnetic resonance imaging (MRI) will be performed to evaluate the presence of Pulmonary Hypertension (PH). The TTEs that were performed by local standards will be collected and undergo central interpretation using European society of Cardiology / European respiratory society (ESC/ERS) guidelines to confirm the local interpretation.
  Interventions: Other: Blood Sample; Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Other: Blood Sample — Blood samples will be taken and analyzed to evaluate the presence of PH.
Diagnostic Test: Cardiac MRI — Cardiac MRI will be performed to evaluate the presence of PH.

SUMMARY:
The primary purpose of this study is to estimate the percentage of participants in the population considered clinically as not having pulmonary hypertension (PH) that are positive for PH biomarker (micro ribonucleic acid [RNA]); estimate the percentage of participants in the population considered clinically as not having PH that are positive for PH by cardiac magnetic resonance imaging (MRI) and compare results of the MRI to the biomarker results; to determine the performance of the biomarker signatures identified in the CIPHER (NAPUH0001) study in terms of sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV), in a population considered clinically as not having PH.

ELIGIBILITY:
Inclusion Criteria:

* Referred for diagnostic work-up for pulmonary hypertension (PH)
* With low or intermediate (but not high) probability of PH by transthoracic echocardiography (TTE) according to European Society of Cardiology (ESC)/ European Respiratory Society (ERS) Guidelines if at the time of enrollment Right Heart Catheterization (RHC) is not deemed to be clinically indicated
* Medically stable on the basis of physical examination, medical history and vital signs performed at screening. Any abnormalities must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and initialed by the investigator
* Must sign an Informed consent (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Must sign a separate approval in the ICF if he or she agrees to provide an optional (DNA) sample for research. Refusal to give consent for the optional (DNA) research sample does not exclude a participant from participation in the study

Exclusion Criteria:

* Undergone RHC within 2 years
* Participants requiring renal dialysis
* Participants post-lung or heart transplant
* Severe left ventricular dysfunction: left ventricular ejection fraction less then (<) 35 percent
* Ongoing Contagious respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants in the Population Considered Clinically as not Having PH that are Positive for PH Biomarker | Up to 90 Days
  Percentage of (transthoracic echocardiography [TTE] low/intermediate probability) participants who are positive for the biomarker will be estimated.
Percentage of Participants Considered Clinically as not Having PH that are Positive for PH by Cardiac MRI | Up to 90 Days
  Percentage of participants considered clinically as not having PH that are positive for PH by cardiac magnetic resonance imaging (MRI) will be evaluated.
Performance of Biomarker Results | Up to 90 Days
  The performance of the biomarker in the diagnosis of PH will be evaluated using the MRI result.
Performance of the Biomarker Signatures Identified in the CIPHER Study in Terms of Sensitivity, specificity, positive predictive value (PPV) and Negative Predictive Value (NPV), in Participants not Having PH | Up to 90 Days
  Performance of the biomarker signatures identified in the CIPHER study in terms of sensitivity, specificity, PPV and NPV, in a population considered clinically as not having PH will be estimated.

SECONDARY OUTCOMES:
Biomarker Data Pooled with the Biomarker Data Collected from the CIPHER (NAPUH0001) Study | Up to 90 Days
  The biomarker data collected from participants with low/intermediate suspicion of PH in the CIPHER-MRI study will be pooled with the data collected from the high to intermediate suspicion of PH participants in the CIPHER (NAPUH0001) study to evaluate the performance of the biomarker signature(s) developed in CIPHER (NAPUH0001).

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (8):
- Germany (3):
  - Universitatsklinikum Bonn, Bonn
  - Universitaetsklinikum Giessen, Giessen
  - Universitatsklinikum Schleswig Holstein, Lübeck
- United Kingdom (5):
  - Royal United Hospital, Bath
  - National Waiting Times Centre Board Golden Jubilee National Hospital, Glasgow
  - Royal Free Hospital, London
  - Hammersmith Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency